CLINICAL TRIAL: NCT00961792
Title: Individual Differences After Consumption of Alcohol and Other Common Substances and Long-Term Follow-Up of Social Drinking, Young Adults
Brief Title: Chicago Social Drinking Project
Acronym: CSDP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 12119a; 5R01AA013746 (NIH)
Record Dates: First submitted 2009-08-11; First posted 2009-08-19 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; trichlorosucrose; Diphenhydramine; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Beverage with Heavy Alcohol Dose (Experimental): Beverage containing 0.8 g/kg alcohol
  Interventions: Drug: Ethanol
- Beverage with Low Alcohol Dose (Experimental): Beverage containing 0.4 g/kg alcohol
  Interventions: Drug: Ethanol
- Beverage with No alcohol (Placebo) (Placebo Comparator): Beverage containing 0.0 g/kg alcohol to act as placebo
  Interventions: Drug: Placebo
- Beverage with Diphenhydramine (Experimental): Beverage containing 1.5 standard dose of Diphenhydramine (Benadryl)
  Interventions: Drug: Diphenhydramine
- Beverage with Caffeine (Experimental): Beverage containing the equivalent of 1.5 times participant's average caffeine consumption
  Interventions: Drug: Caffeine
- Beverage in Natural Environment (No Intervention): Participant consumes alcohol containing beverages or non-alcohol beverages in natural environment

INTERVENTIONS:
Drug: Ethanol — Beverage containing 0.8 g/kg ethanol, 0.4 g/kg ethanol
  Other Names: Kool-Aid; Splenda; Everclear
  Arms: Beverage with Heavy Alcohol Dose; Beverage with Low Alcohol Dose
Drug: Placebo — Beverage containing 0.0 g/kg alcohol to act as placebo
  Arms: Beverage with No alcohol (Placebo)
Drug: Diphenhydramine — Beverage containing dose equivalent to 1.5 standard doses of Diphenhydramine (Benadryl)
  Other Names: Benadryl
  Arms: Beverage with Diphenhydramine
Drug: Caffeine — Beverage containing the equivalent of 1.5 times the participant's daily caffeine intake
  Arms: Beverage with Caffeine

SUMMARY:
This study attempts to elucidate the factors that contribute to escalation and maintenance of excessive ethanol drinking in young adults by:

1. Examining subjective and objective response differences to alcohol and other common substances in a sample of adults with varying consumption patterns.
2. Determining whether response to alcohol and other substances is predictive of future consumption patterns through longitudinal follow-up interviews.
3. Examining the relationship between responses to alcohol and other substances at baseline and re-examination testing to evaluate if consumption patterns moderate this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Weigh between 110-210 lbs
* Drink alcohol at least once weekly with weekly "binge" drinking episodes
* Available to complete in-person screening and 2, 4 hour experimental sessions at the University of Chicago
* Available by phone, mail, or Internet for follow-up interviews for at least 2 years following sessions

Exclusion Criteria:

* Current or past major medical or psychiatric disorders including alcohol and substance dependence

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-03; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Subjective response to alcohol and other common substances utilizing mood questionnaires in adult drinkers | Measured during 5 timepoints at each experimental session: 1) Pre-drink baseline, 2) +30 minutes, 3) +60 minutes, 4) +120 minutes, and 5) +180 minutes following the initiation of beverage consumption

SECONDARY OUTCOMES:
Substance Use Behavior Reported During Follow-Up Interviews | Measured at 3, 6, 9, 12, 15, 18, 21, 24, 36, 48, and 60 months following the final experimental session

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C King, PhD, Principal Investigator — University of Chicago
Locations (1):
- Clinical Addictions Research Laboratory, Chicago, Illinois, United States

REFERENCES:
- [Background] King AC, Byars JA. Alcohol-induced performance impairment in heavy episodic and light social drinkers. J Stud Alcohol. 2004 Jan;65(1):27-36. doi: 10.15288/jsa.2004.65.27. PMID 15000501
- [Background] King AC, Houle T, de Wit H, Holdstock L, Schuster A. Biphasic alcohol response differs in heavy versus light drinkers. Alcohol Clin Exp Res. 2002 Jun;26(6):827-35. PMID 12068251
- [Result] Rueger SY, McNamara PJ, King AC. Expanding the utility of the Biphasic Alcohol Effects Scale (BAES) and initial psychometric support for the Brief-BAES (B-BAES). Alcohol Clin Exp Res. 2009 May;33(5):916-24. doi: 10.1111/j.1530-0277.2009.00914.x. Epub 2009 Mar 11. PMID 19320625
- [Result] Epstein AM, Sher TG, Young MA, King AC. Tobacco chippers show robust increases in smoking urge after alcohol consumption. Psychopharmacology (Berl). 2007 Feb;190(3):321-9. doi: 10.1007/s00213-006-0438-8. Epub 2006 Jun 28. PMID 16804691
- [Result] Brumback T, Cao D, King A. Effects of alcohol on psychomotor performance and perceived impairment in heavy binge social drinkers. Drug Alcohol Depend. 2007 Nov 2;91(1):10-7. doi: 10.1016/j.drugalcdep.2007.04.013. Epub 2007 Jun 8. PMID 17560739
- [Result] King A, Epstein A, Conrad M, McNamara P, Cao D. Sex differences in the relationship between alcohol-associated smoking urge and behavior: a pilot study. Am J Addict. 2008 Sep-Oct;17(5):347-53. doi: 10.1080/10550490802268140. PMID 18770076
- [Result] King AC, Epstein AM. Alcohol dose-dependent increases in smoking urge in light smokers. Alcohol Clin Exp Res. 2005 Apr;29(4):547-52. doi: 10.1097/01.alc.0000158839.65251.fe. PMID 15834219
- [Result] King A, Vena A, Hasin DS, deWit H, O'Connor SJ, Cao D. Subjective Responses to Alcohol in the Development and Maintenance of Alcohol Use Disorder. Am J Psychiatry. 2021 Jun;178(6):560-571. doi: 10.1176/appi.ajp.2020.20030247. Epub 2021 Jan 5. PMID 33397141
- [Derived] King AC, Cao D, deWit H, O'Connor SJ, Hasin DS. The role of alcohol response phenotypes in the risk for alcohol use disorder. BJPsych Open. 2019 Apr 22;5(3):e38. doi: 10.1192/bjo.2019.18. PMID 31685074
- [Derived] King AC, Hasin D, O'Connor SJ, McNamara PJ, Cao D. A Prospective 5-Year Re-examination of Alcohol Response in Heavy Drinkers Progressing in Alcohol Use Disorder. Biol Psychiatry. 2016 Mar 15;79(6):489-98. doi: 10.1016/j.biopsych.2015.05.007. Epub 2015 May 14. PMID 26117308
- [Derived] King AC, McNamara PJ, Hasin DS, Cao D. Alcohol challenge responses predict future alcohol use disorder symptoms: a 6-year prospective study. Biol Psychiatry. 2014 May 15;75(10):798-806. doi: 10.1016/j.biopsych.2013.08.001. Epub 2013 Oct 2. PMID 24094754
- [Derived] King AC, de Wit H, McNamara PJ, Cao D. Rewarding, stimulant, and sedative alcohol responses and relationship to future binge drinking. Arch Gen Psychiatry. 2011 Apr;68(4):389-99. doi: 10.1001/archgenpsychiatry.2011.26. PMID 21464363
- See also: Study Website — https://socialdrinking.bsd.uchicago.edu/